CLINICAL TRIAL: NCT04998253
Title: A Randomized Pilot Clinical Trial of the Effects in Oxygenation and Hypoxic Pulmonary Vasoconstriction of Sevoflurane in Patient's Whit ARDS Secondary to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV2)
Brief Title: Effects in Oxygenation and Hypoxic Pulmonary Vasoconstriction in ARDS Secondary to SARS-CoV2
Acronym: COVID-19
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Unidad Temporal COVID-19 en Centro Citibanamex (Other)
Responsible Party: Principal Investigator, Adrian Palacios-Chavarria, MD, Principal investigator, Unidad Temporal COVID-19 en Centro Citibanamex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-CIE-011-20160627
Record Dates: First submitted 2021-05-19; First posted 2021-08-10 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Hypoxic Pulmonary Vasoconstriction; Hypoxemia; Acute Respiratory Distress Syndrome; SARS-CoV-2 Acute Respiratory Disease
MeSH Terms: conditions — Hypoxia; Respiratory Distress Syndrome | interventions — Treatment Outcome; Ferritins

STUDY DESIGN:
Intervention Model Description: Target Population: Patients with ARDS secondary to COVID-19 on invasive mechanical ventilation.
  Accessible population: Patients with ARDS secondary to COVID-19 on invasive mechanical ventilation admitted to the Temporary COVID-19 Citibanamex Unit.
  7.3 Randomization Simple randomization will be carried out using an envelope containing each sedative with 2 treatment groups. Taking into account 5% losses, by the formula: Sample adjusted to losses = n (1/1 - R) n = number of subjects without losses R = expected proportion of losses A person outside the study will place the indicated therapy inside identical opaque envelopes numbered 1 to 82 and then in a closed box. We will use the envelopes consecutively with the indicated therapy. Neither the researcher nor the people related to the study or the treatment will know the therapy that each patient will receive.
Who Masked: Care Provider
Masking Description: A person outside the research group will randomize the patients through the simple selection of the two drugs, once their admission to the intensive care unit is requested. We will not carry out the blinding of the researchers since the use of sevoflurane requires an external computer that cannot be replicated for the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Sevofruorane (Svofast) (Experimental): Experimental group: will receive sedation with sevoflurane with an infusion rate to maintain MAC of 0.7 and fentanyl 1mcg /kg/hour.
  Inhalation sedation The AnaConda device (Sedana Medical, Ireland) is placed between the endotracheal tube and the ventilator circuit. The anesthetic infusion line is attached to a syringe, from where the anesthetic (sevoflurane) will be delivered to said device. The sample line will be taken to the anesthetic gas analyzer whit the Carescape B450 multiparametric monitors (General Electric, Finland) for MAC control. The anesthetic gas outlet port will be attached to the absorbent material container.
  Interventions: Drug: Effects in oxygenation and hypoxic pulmonary vasoconstriction
- Group 2: Propofol (Diprivant) (Active Comparator): Control group: will receive sedation with Propofol (Diprivant) at doses of 20-50mcg/kg/min and fentanyl (Fentanest) at doses of 1 to 2mcg/kg /hour.
  For both groups, the doses will be titrated to maintain a RASS score between -3 to -4 in both groups.
  Both groups will receive cisatracurium (Nimbex) as a continuous infusion of 3 to 5mcg / kg/min for 48 hours. We will maintain sedation for both groups with the same scheme for 48 hours, after which the drugs used for sedation will be modified at the discretion of the intensive care physicians.
  Interventions: Drug: Effects in oxygenation and hypoxic pulmonary vasoconstriction

INTERVENTIONS:
Drug: Effects in oxygenation and hypoxic pulmonary vasoconstriction — Determination of the anti-inflammatory effect. The anti-inflammatory effect is assessed with serum measurement of interleukin 6 (IL-6), C-reactive protein (CRP), ferritin, DHL (lactic dehydrogenase), taken by venipuncture on admission, at 24 and 48 hours.
  The following measurements will be performed: pulmonary artery systolic and diastolic pressure (PASP, PADP respectively), central venous pressure (CVP), pulmonary artery occlusion pressure (PAOP), pulmonary vascular resistance (PVR), systemic vascular resistance (SVR), right ventricular stroke work (RVSW) and left ventricular work (LVSW). Stroke volume (and cardiac output) will be computed using the thermodilution technique averaging three consecutive injections with 10 ml of 0.9% saline solution.
  Other Names: 3. Compare anti-inflammatory effect (determined by serum levels of IL-6, CRP, ferritin, DHL) of sevoflurane against propofol.; 1. Compare the effect on the pulmonary circulation of sevoflurane against Propofol.

SUMMARY:
Summary Currently, the COVID-19 pandemic has overtaken health systems worldwide, exceeding the capacity of intensive care units. In addition to this, countries such as the United States have reported a decrease in the supplies of drugs such as Propofol and Midazolam (traditionally used as sedatives in patients with invasive mechanical ventilation), so in the absence until now of a specific treatment against SARS-COV-2 virus, improving the support strategies in patients in the severe spectrum of the disease Acute Respiratory Distress Syndrome (ARDS) is a priority.

Given the global state of emergency due to COVID-19, the use of sevoflurane has the potential to mitigate the shortages of sedative drugs, promote the recovery of patients with ARDS, and potentially reduce mortality.

A study will be conducted to evaluate the effect of sevoflurane as inhalation sedation in patients with ARDS secondary to SARS-COV2 compared to the standard. The primary objective of the study is to assess the difference in oxygenation, for which the calculation of the partial pressure of arterial oxygen to fractional inspired oxygen concentration ratio (PaO2 / FiO2) will be used at 24 and 48 hours. Also, the effect of the possible attenuation or inhibition of hypoxic pulmonary vasoconstriction will be evaluated by hemodynamic monitoring with a pulmonary artery catheter and transthoracic echocardiography and its possible effect on the right ventricle.

Outcome: we expect an improvement in oxygenation and consequently a reduction in the days of invasive mechanical ventilation, stay in the intensive care unit (ICU) and hospital. In addition to evaluating its possible anti-inflammatory effect and probably establishing a safe and effective alternative and possibly with greater benefits compared to standard intravenous sedation.

DETAILED DESCRIPTION:
1. Background.

   The lung is the main organ affected in the SARS-COV-2 virus infection, in an observational study, it was reported that up to 42% of patients developed ARDS and of these, up to 81% required intensive care treatment. The mortality reported at the beginning of the pandemic for patients with ARDS secondary to COVID-19 was close to 90%, however, a recent study places mortality at 32%, a figure that is related to that reported for ARDS of other etiologies.

   To date, few interventions have been shown to have an impact on the mortality of patients with ARDS (of any etiology) in mechanical ventilation: judicious use of PEEP (pressure at the end of expiration), ventilation with low tidal volume (6 ml/kg predicted weight), limit plateau pressure (Pplt) to less than 30 cmH2O, maintain alveolar conduction pressure (DP) <15cmH2O and early use of ventilation in the prone position.

   The use of alveolar recruitment maneuvers and neuromuscular blockade, although controversial, are widely used with variable impact on mortality. The use of VV ECMO (Veno-venous configuration extracorporeal oxygenation membrane), ECCO2R (extracorporeal carbon dioxide removal), and NO (nitric oxide) systems are limited by availability and high cost with inconsistent results in mortality in ARDS.

   Therefore, the search for other cost-effective strategies for the treatment of ARDS has led to the consideration in recent years of the use of other drugs such as volatile anesthetics.

   Jabaudon et al. conducted a study of sedation with sevoflurane in patients with ARDS where they documented an improvement in the PaO2/FiO2 ratio in the first two days compared with patients sedated with midazolam. It should be clarified that the study showed no difference in mortality between the two groups however this can be attributed to the number of subjects included (n = 50).

   Sevoflurane offers several advantages as a sedative agent in ARDS patients on mechanical ventilation. They depress the ventilatory response to hypoxia and hypercapnia with a dose and time-dependent effect. The response to hypoxia is altered from 0.1 MAC (minimum alveolar concentration) of the halogenated agent and disappears above 1.1 MAC, with moderate effects on hypercapnia. It is a potent bronchodilator that potentiates the effect of neuromuscular blockers and has cardioprotective properties.

   However, there are potential disadvantages of sevoflurane, depression of cardiac contractile function has been observed in animal models, as well as dose-dependent lusitropic alteration, and inhibition of the mechanisms that facilitate hypoxic pulmonary vasoconstriction (HPV).

   Currently, anti-inflammatory properties of sevoflurane have been documented in animal models with ARDS, with a significant reduction of cytokines such as IL-1b (interleukin 1 beta), IL-6, IL-10, TNFa (tumor necrosis factor-alpha), TGF- b (transforming growth factor-beta) among others. These findings were also corroborated in humans by Jabaudon et al.
2. Justification. Currently, the COVID-19 pandemic has overtaken health systems worldwide, exceeding the capacity of intensive care units. In addition to this, countries such as the United States have reported a decrease in the supplies of drugs such as Propofol and Midazolam (traditionally used as sedatives in patients with invasive mechanical ventilation), so in the absence until now of a specific treatment against SARS-COV-2 virus [36], improving the support strategies in patients in the severe spectrum of the disease (ARDS) is a priority.
3. Statement of the Problem. Experimental evidence in animal models and with humans reveal the anti-inflammatory effect of sevoflurane at the pulmonary level with improvement in oxygenation in the setting of adult respiratory distress syndrome regardless of its etiology.

   Given the global state of emergency due to COVID-19, the use of sevoflurane has the potential to mitigate the shortages of sedative drugs, promote the recovery of patients with ARDS, and potentially reduce mortality.

   Therefore, it is relevant to define the effect of sevoflurane on cardiac function, especially on the right ventricle, as well as its ability to attenuate the hypoxic vasoconstriction mechanism, since it would allow establishing its risk profile in this population and standardizing its use.
4. Research Question. Can sevoflurane improve oxygenation in patients with ARDS secondary to COVID-19 without significantly affecting the mechanism of hypoxic vasoconstriction or right ventricular function?
5. Primary objective. To determine whether sedation with sevoflurane improves oxygenation without producing significant changes in the mechanism of hypoxic vasoconstriction (determined by changes in pulmonary vascular resistance) or in right ventricular function.

   5.1 Secondary objectives: Compare the effect on the pulmonary circulation of sevoflurane against Propofol.

   Compare the effect on the right ventricular function of sevoflurane versus Propofol.

   Compare anti-inflammatory effect (determined by serum levels of IL-6, CRP, ferritin, DHL) of sevoflurane against propofol.
6. Hypothesis. Sevoflurane improves oxygenation in patients with ARDS secondary to COVID-19 without a significant impact on the mechanism of HVP and right ventricular function.
7. Patients and Methods.

   7.1 Randomization Simple randomization will be carried out using an envelope containing each sedative with 2 treatment groups, in total 11 patients will be placed in each group. Considering 5% losses, by the formula: Sample adjusted to losses = n (1/1 - R) n = number of subjects without losses R = expected proportion of losses A person outside the study will place the indicated therapy inside identical opaque envelopes numbered 1 to 22 and then in a closed box. The investigators will use the envelopes consecutively with the indicated therapy. Neither the researcher nor the people related to the study or the treatment will know the therapy that each patient will receive.

   7.2 Sample calculation: The investigators based the sample calculation on the article published by Jabaudon and collaborators.

   Using the formula for the difference of means: (Alpha). Sample size estimation for two tails n=((Z1-β±Z1-α/2)2*σ)/((µ0-µ1))

   Where:

   Zα = value of z related to α = 0.05 (extracted from reference tables) Zβ = value of z related to β = 0.20 (power of 80%). SD = standard deviation μ0 = group A mean µ1 = mean of group B

   According to the example, substituting the values. It would be as follows:

   Zα = 1.96 Zβ = -0.84 SD = 2 µ0 = 205 ± 56 μ1 = 166 ± 59

   It is necessary to include 39 patients in each group if it is desired to obtain 80% statistical power with an error α of 0.05. If it is desired to achieve greater power, i.e. 99% with an error α of 0.01, 107 should be included per group. To detect a mean difference of -141, seeking to achieve that with the use of sevoflurane oxygenation improves by using the PaO2/FIO2 ratio.

   8.1 Randomization. A person outside the research group will randomize the patients through the simple selection of the two drugs, once their admission to the intensive care unit is requested. The investigators will not carry out the blinding of the researchers since the use of sevoflurane requires an external computer that cannot be replicated for the control group.

   8.2 Definition of the maneuver to be performed. Experimental group: will receive sedation with sevoflurane with an infusion rate to maintain MAC of 0.7 and fentanyl 1mcg /kg/hour Control group: will receive sedation with Propofol at doses of 20-50mcg/kg/min and fentanyl at doses of 1 to 2mcg/kg /hour.

   For both groups, the doses will be titrated to maintain a RASS score between -3 to -4 in both groups.

   Both groups will receive cisatracurium as a continuous infusion of 3 to 5mcg / kg/min for 48 hours. The investigators will maintain sedation for both groups with the same scheme for 48 hours, after which the drugs used for sedation will be modified at the discretion of the intensive care physicians.

   8.2 Evaluation of Oxygenation. The primary objective of the study is to assess the difference in oxygenation in both groups, for which the calculation of the PaO2 / FiO2 ratio will be used, taking peripheral arterial blood, with FiO2 at 100% one hour after the start of sedation corresponding to each group, again at 24 and 48 hours.

   8.3 Effect on the mechanism of hypoxic pulmonary vasoconstriction.

   Hypoxic pulmonary vasoconstriction (HPV) is a complex mechanism that responds to local effects on oxygen depletion probably through precapillary alveolar vasoconstriction mediated by intrinsic, sympathetic, and perhaps other humoral agents. Due to the difficulty of studying this mechanism, the investigators will use surrogate methods. For this purpose, the use of pulmonary vascular resistance is considered, which will represent changes in pulmonary vascular tone and will be determined invasively through a pulmonary arterial catheter (Swan-Ganz) for which the following formula will be used:

   PVR=(MPAP-LAP)/CO Where PVR = pulmonary vascular resistance, MPAP = mean pulmonary artery pressure, LAP = left atrial pressure or pulmonary wedge pressure and CO = cardiac output.

   The research group agreed to calculate the PVR using parameters obtained by the Swan-Ganz catheter because it is the gold standard for the study of pulmonary circulation.

   Another surrogate method will be the shunt fraction, for which mixed venous blood (taken from the pulmonary artery) and systemic arterial blood (taken from the radial artery) with a FiO2 (inspired oxygen fraction) of 100% will be used. Alterations in the hypoxic vasoconstriction mechanism will be reflected as an increase or decrease in the short-circuit fraction, for the above, the following formula will be applied:

   SCF=(CcO2-CaO2)/(CcO2-CvO2) Where SF = Shunt fraction, CcO2 = capillary oxygen content, CaO2 = arterial oxygen content and CvO2 = venous oxygen content.

   CcO2=1.34xHbx1+0.0031xPaO2 Where Hb = Hb concentration in g / dL, 1 represents 100% saturation of hemoglobin at the level of the alveolar capillaries, 0.0031 is the oxygen dilution constant in plasma and PaO2 is the peripheral arterial oxygen partial pressure in mmHg.

   CaO2=1.34xHbxSaO2+0.0031xPaO2 Where SaO2 is the peripheral arterial oxygen saturation (numerical value) and paO2 is the peripheral arterial oxygen partial pressure in mmHg.

   CvO2=1.34xHbxSvO2+0.0031xPvO2 Where SvO2 is the mixed venous oxygen saturation (numerical value) and PvO2 is the partial pressure of oxygen at the venous level.

   The shunt fraction was considered by the research group as another surrogate to evaluate the phenomenon of hypoxemic pulmonary vasoconstriction, the inhibition of this would produce an increase in the shunt fraction by allowing blood circulation through non-ventilated alveoli. The shunt fraction will be recorded one hour after the start of sedation corresponding to each group, again at 24 and 48 hours.

   8.4 Evaluation of right ventricular function. The investigators will assess the right ventricular function by determining invasive parameters of the pulmonary artery catheter. The investigators will measure parameters one hour after the start of sedation for each group, again at 24 and 48 hours.

   8.5 Determination of the anti-inflammatory effect. The anti-inflammatory effect is assessed with serum measurement of interleukin 6 (IL-6), C-reactive protein (CRP), ferritin, DHL (lactic dehydrogenase), taken by venipuncture on admission, at 24 and 48 hours.

   8.6 Measurement of dead space (DS). Quantitative lateral flow capnography will be performed through a Carescape B450 multiparametric (General Electric, Finland).

   The physiological dead space expressed as a percentage will be calculated using the Bohr formula:

   DS=(PACO2-PEtCO2)/PACO2 Where DS = dead space, PaCO2 = partial pressure of arterial CO2 in mmHg, PEtCO2 = end tidal CO2 pressure in mmHg.

   Measurements will be made one hour after the start of sedation for each group, again at 24 and 48 hours.

   8.7 Alveolar ventilation monitoring.

   The investigators will measure the partial pressure of CO2 at the peripheral arterial blood and the values will be recorded after the start of sedation corresponding to each group, as well as at 24 and 48 hours.

   8.8 Mechanical Ventilation.

   Mechanical ventilation will be carried out with Mindray SV300 ventilators (Mindray, China) for the case of the control groups, in the case of the experimental group, due to the type of connection required for the activated carbon filter, Avea ventilators (Carefusion, United States) will be used or Dräger Evita Infinity V500 (Dräger, Germany).

   After intubation, the investigators will perform a staircase recruitment maneuver.

   8.8.1 Staircase recruitment maneuver.

   Pressure assist-control mode will be programmed with an inspiratory pressure of 15 cm H2O, respiratory rate of 10 breaths per minute, inspiration-expiration ratio (IRR) 1: 1, FiO2 100% and PEEP of 25 cm H2O for 1 minute, then PEEP will be increased to 30 cmH2O for 1 minute and finally, PEEP will increase to 35 cm H2O for 1 minute.

   8.8.2 PEEP titration.

   After the alveolar recruitment maneuver, PEEP will be titrated based on the best compliance (descending fashion).

   In assist-control mode by volume with decelerated flow (not all the ventilators used to offer a continuous flow option), a volume of 6ml / kg of predicted weight will be programmed with the following formula:

   Men = 50 + [0.91 x (size in cm-152.4)] Women = 45.5 + [0.91 x (size in cm-152.4)]

   The respiratory rate will be programmed at 20 breaths per minute with 1: 2 inspiration: expiration (IRR) ratio, FiO2 100%, PEEP of 23cmH2O. The selected PEEP will be maintained for 1 minute and lung compliance will be measured with an inspiratory pause of 3 seconds, which will be recorded, a total of 3 minutes will be completed with the selected PEEP after which 3cmH2O will be decreased, repeating this process until the best distensibility is obtained. The best static compliance, which will be recorded and the PEEP will be programmed 2cmH2O over the PEEP in which the best compliance has been obtained. Once the PEEP has been titrated, it will not be modified within 48 hours, unless airway pressure targets are not maintained (alveolar conduction pressure or plateau pressure).

   8.8.3 Objectives of mechanical ventilation: Tidal volume ventilation calculated at 6ml / kg predicted weight. Plateau pressure = or <27 cmH2O Alveolar conduction pressure = or <14 cmH2O FiO2 to maintain SpO2 between 92 to 94% Arterial pH> 7.25. Minimize Auto-PEEP 3.8.4 Measurements of lung mechanics and ventilation parameters.

   The following measurements will be made through the ventilator software tools:

   Plateau pressure (Pplt) by applying a 3-second inspiratory pause.

   Alveolar driving pressure (DP): using the following formula:

   DP=Pplt-PEEP

   Static compliance (Cest) = by the following formula:

   Cest=Tidal Volume/DP Airway resistance (Raw), which will be calculated using the following formula. RVA=(Ppk-Pplt)/Flow Where Ppk is the peak pressure, Pplt is the plateau pressure, and flow is the volume that enters the system during inspiration in one second.

   The investigators will record the minute volume and respiratory rate.

   The investigators will record the measurement of Dp, Cest, and Pplt 1 hour after the start of the corresponding sedation and again at 24 and 48 hours.

   The investigators will document the average minute volume and respiratory rate on days 1 and 2.

   8.8.5 Ventilation in the prone position.

   Patients who, after 24 hours of the recruitment and PEEP titration maneuver, have a PaO2 / FiO2 ratio <150mmHg will be candidates for ventilation in the prone position.

   8.9 Inhalation sedation The AnaConda device (Sedana Medical, Ireland) is placed between the endotracheal tube and the ventilator circuit. The anesthetic infusion line is attached to a syringe, from where the anesthetic (sevoflurane) will be delivered to said device. The sample line will be taken to the anesthetic gas analyzer for MAC control (End-expiratory concentration "EEC" of the anesthetic). The anesthetic gas outlet port will be attached to the absorbent material container.

   Filling the syringe and purging the infusion line: the infusion lines and sampling line must be supplied by the manufacturer AnaConda since volatile anesthetics can dissolve plastic materials. The syringes must be filled with the special adapter which is placed on the anesthetic bottle, avoiding leaks to avoid environmental contamination. Since the infusion line has a dead space of 1.2 ml in volume, a bolus will be programmed in the infusion pump. Once the line has been purged, the infusion rate will be adjusted to the minute volume or MAC of the anesthetic. The rate will be between 2 to 10 ml/hour or until obtaining a MAC 0.7.

   Unwanted effects with the use of AnaConda:

   Increased dead space (approximately 100 ml) Hemodynamic effects in case of overdose. Effects of sevoflurane administration Drug Interactions with Sevoflurane. There is no evidence of interaction with other drugs other than those indicated by the anesthetic technical datasheet.

   8.10 Hemodynamic monitoring and pressure recording. Carescape B450 multiparametric monitors (General Electric, Finland) will be used for the measurement and recording of pressures, as well as standard transducers for the measurement of invasive pressures.

   A central venous catheter (triple-lumen) of 7 Fr and 20 cm in length (Teleflex, USA) will be installed for all patients through left internal jugular access, as well as a 7 Fr Swan-Ganz type pulmonary artery catheter and 110 cm (Edwards Lifesciences, USA) using 11 cm long 8 Fr percutaneous introducers (Teleflex, USA) through the right internal jugular vein.

   For venous cannulation, a modified Seldinger technique will be used with ultrasound guidance with a 5-10 MHz linear transducer L-38 (Fujifilm Sonosite Europe, The Netherlands) with a Sonosite SII ultrasound device (Fujifilm Sonosite Europe, The Netherlands). After the placement of the venous catheters, a portable chest X-ray will be taken to confirm that these catheters have the usual position and rule out complications.

   The following measurements will be performed: pulmonary artery systolic and diastolic pressure (PASP, PADP respectively), central venous pressure (CVP), pulmonary artery occlusion pressure (PAOP), pulmonary vascular resistance (PVR), systemic vascular resistance (SVR), right ventricular stroke work (RVSW) and left ventricular work (LVSW). Stroke volume (and cardiac output) will be computed using the thermodilution technique averaging three consecutive injections with 10 ml of 0.9% saline solution.

   Measurements will be made by two operators and will be recorded one hour after the start of sedation for each group and at 24 and 48 hours. In the case of systolic, diastolic, and mean pressure, the averages at 24 and 48 hours will be recorded.

   The record will be made one hour after the start of the sedation assigned to each group, at 24 and 48 hours after the averages of the mean systemic arterial pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years
2. Both genders
3. Diagnosis of COVID-19 (SARS-COV2) with moderate to severe ARDS from the Berlin classification (PaO2 / FiO2: < 200).

Exclusion Criteria:

1. Acute kidney failure.
2. Severe liver failure
3. Suspected or documented intracranial hypertension.
4. Family history of malignant hyperthermia.
5. History of malignant hyperthermia.
6. Documented chronic lung disease.
7. Documented chronic pulmonary hypertension
8. Patients who do not sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Oxygenation | 24 and 48 hours
  The primary objective of the study is measure the difference in the oxygenation whit two different methods of sedation, inhaled (sevorane) and intravenous (propofol). The oxygenation will be measured whit PaO2 / FiO2 ratio will be used, taking peripheral arterial blood, with FiO2 at 100% one hour after the started of sedation corresponding to each group, again at 24 and 48 hours.
The effect in the hypoxic pulmonary vasoconstriction whit two different type sedation. | 24 and 48 hours
  The changes in pulmonary vascular tone and will be measured invasively through a pulmonary arterial catheter (Swan-Ganz) for which the following formula will be used:
  PVR=(MPAP-LAP)/CO Where PVR = pulmonary vascular resistance (dyn*s/cm), MPAP = mean pulmonary artery pressure (mm Hg), LAP = left atrial pressure or pulmonary wedge pressure (mm Hg) and CO = cardiac output (L/min). *79.92 is a constant to equal the units.

SECONDARY OUTCOMES:
Determination of the anti-inflammatory effect. | 24 and 48 hours
  The anti-inflammatory effect will be measured with serum levels of interleukin 6 (IL-6), C-reactive protein (CRP), ferritin, DHL (lactic dehydrogenase), taken by venipuncture on admission, at 24 and 48 hours.
Measurement of dead space. | 24 and 48 hours
  The physiological dead space expressed as a percentage will be calculated using the Bohr formula:
  DS=(PACO2-PEtCO2)/PACO2 Where DS = dead space, PaCO2 = partial pressure of arterial CO2 in mmHg, PEtCO2 = end tidal CO2 pressure in mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Adrián Palacios Chavarria, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ge H, Wang X, Yuan X, Xiao G, Wang C, Deng T, Yuan Q, Xiao X. The epidemiology and clinical information about COVID-19. Eur J Clin Microbiol Infect Dis. 2020 Jun;39(6):1011-1019. doi: 10.1007/s10096-020-03874-z. Epub 2020 Apr 14. PMID 32291542
- [Result] Lu R, Zhao X, Li J, Niu P, Yang B, Wu H, Wang W, Song H, Huang B, Zhu N, Bi Y, Ma X, Zhan F, Wang L, Hu T, Zhou H, Hu Z, Zhou W, Zhao L, Chen J, Meng Y, Wang J, Lin Y, Yuan J, Xie Z, Ma J, Liu WJ, Wang D, Xu W, Holmes EC, Gao GF, Wu G, Chen W, Shi W, Tan W. Genomic characterisation and epidemiology of 2019 novel coronavirus: implications for virus origins and receptor binding. Lancet. 2020 Feb 22;395(10224):565-574. doi: 10.1016/S0140-6736(20)30251-8. Epub 2020 Jan 30. PMID 32007145
- [Result] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Result] Ferrando C, Suarez-Sipmann F, Mellado-Artigas R, Hernandez M, Gea A, Arruti E, Aldecoa C, Martinez-Palli G, Martinez-Gonzalez MA, Slutsky AS, Villar J; COVID-19 Spanish ICU Network. Clinical features, ventilatory management, and outcome of ARDS caused by COVID-19 are similar to other causes of ARDS. Intensive Care Med. 2020 Dec;46(12):2200-2211. doi: 10.1007/s00134-020-06192-2. Epub 2020 Jul 29. PMID 32728965
- [Result] Brochard L, Slutsky A, Pesenti A. Mechanical Ventilation to Minimize Progression of Lung Injury in Acute Respiratory Failure. Am J Respir Crit Care Med. 2017 Feb 15;195(4):438-442. doi: 10.1164/rccm.201605-1081CP. PMID 27626833
- [Result] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Result] Amato MB, Barbas CS, Medeiros DM, Magaldi RB, Schettino GP, Lorenzi-Filho G, Kairalla RA, Deheinzelin D, Munoz C, Oliveira R, Takagaki TY, Carvalho CR. Effect of a protective-ventilation strategy on mortality in the acute respiratory distress syndrome. N Engl J Med. 1998 Feb 5;338(6):347-54. doi: 10.1056/NEJM199802053380602. PMID 9449727
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Brower RG, Lanken PN, MacIntyre N, Matthay MA, Morris A, Ancukiewicz M, Schoenfeld D, Thompson BT; National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med. 2004 Jul 22;351(4):327-36. doi: 10.1056/NEJMoa032193. PMID 15269312
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Result] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Result] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Moss M, Huang DT, Brower RG, Ferguson ND, Ginde AA, Gong MN, Grissom CK, Gundel S, Hayden D, Hite RD, Hou PC, Hough CL, Iwashyna TJ, Khan A, Liu KD, Talmor D, Thompson BT, Ulysse CA, Yealy DM, Angus DC. Early Neuromuscular Blockade in the Acute Respiratory Distress Syndrome. N Engl J Med. 2019 May 23;380(21):1997-2008. doi: 10.1056/NEJMoa1901686. Epub 2019 May 19. PMID 31112383
- [Result] Combes A, Hajage D, Capellier G, Demoule A, Lavoue S, Guervilly C, Da Silva D, Zafrani L, Tirot P, Veber B, Maury E, Levy B, Cohen Y, Richard C, Kalfon P, Bouadma L, Mehdaoui H, Beduneau G, Lebreton G, Brochard L, Ferguson ND, Fan E, Slutsky AS, Brodie D, Mercat A; EOLIA Trial Group, REVA, and ECMONet. Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome. N Engl J Med. 2018 May 24;378(21):1965-1975. doi: 10.1056/NEJMoa1800385. PMID 29791822
- [Result] Jabaudon M, Boucher P, Imhoff E, Chabanne R, Faure JS, Roszyk L, Thibault S, Blondonnet R, Clairefond G, Guerin R, Perbet S, Cayot S, Godet T, Pereira B, Sapin V, Bazin JE, Futier E, Constantin JM. Sevoflurane for Sedation in Acute Respiratory Distress Syndrome. A Randomized Controlled Pilot Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):792-800. doi: 10.1164/rccm.201604-0686OC. PMID 27611637
- [Result] Patel SS, Goa KL. Sevoflurane. A review of its pharmacodynamic and pharmacokinetic properties and its clinical use in general anaesthesia. Drugs. 1996 Apr;51(4):658-700. doi: 10.2165/00003495-199651040-00009. PMID 8706599
- [Result] Harkin CP, Pagel PS, Kersten JR, Hettrick DA, Warltier DC. Direct negative inotropic and lusitropic effects of sevoflurane. Anesthesiology. 1994 Jul;81(1):156-67. doi: 10.1097/00000542-199407000-00022. PMID 8042785
- [Result] Kerbaul F, Bellezza M, Mekkaoui C, Feier H, Guidon C, Gouvernet J, Rolland PH, Gouin F, Mesana T, Collart F. Sevoflurane alters right ventricular performance but not pulmonary vascular resistance in acutely instrumented anesthetized pigs. J Cardiothorac Vasc Anesth. 2006 Apr;20(2):209-16. doi: 10.1053/j.jvca.2005.05.017. Epub 2006 Jan 19. PMID 16616661
- [Result] Ishibe Y, Gui X, Uno H, Shiokawa Y, Umeda T, Suekane K. Effect of sevoflurane on hypoxic pulmonary vasoconstriction in the perfused rabbit lung. Anesthesiology. 1993 Dec;79(6):1348-53. doi: 10.1097/00000542-199312000-00026. PMID 8267210
- [Result] Ryan D, Frohlich S, McLoughlin P. Pulmonary vascular dysfunction in ARDS. Ann Intensive Care. 2014 Aug 22;4:28. doi: 10.1186/s13613-014-0028-6. eCollection 2014. PMID 25593744
- [Result] Kerbaul F, Bellezza M, Guidon C, Roussel L, Imbert M, Carpentier JP, Auffray JP. Effects of sevoflurane on hypoxic pulmonary vasoconstriction in anaesthetized piglets. Br J Anaesth. 2000 Sep;85(3):440-5. doi: 10.1093/bja/85.3.440. PMID 11103187
- [Result] Lesitsky MA, Davis S, Murray PA. Preservation of hypoxic pulmonary vasoconstriction during sevoflurane and desflurane anesthesia compared to the conscious state in chronically instrumented dogs. Anesthesiology. 1998 Dec;89(6):1501-8. doi: 10.1097/00000542-199812000-00029. PMID 9856726
- [Result] Beck DH, Doepfmer UR, Sinemus C, Bloch A, Schenk MR, Kox WJ. Effects of sevoflurane and propofol on pulmonary shunt fraction during one-lung ventilation for thoracic surgery. Br J Anaesth. 2001 Jan;86(1):38-43. doi: 10.1093/bja/86.1.38. PMID 11575407
- [Result] Matsuse S, Hara Y, Ohkura T. The possible influence of pulmonary arterio-venous shunt and hypoxic pulmonary vasoconstriction on arterial sevoflurane concentration during one-lung ventilation. Anesth Analg. 2011 Feb;112(2):345-8. doi: 10.1213/ANE.0b013e3182025c8e. Epub 2010 Nov 16. PMID 21081765
- [Result] Abe K, Shimizu T, Takashina M, Shiozaki H, Yoshiya I. The effects of propofol, isoflurane, and sevoflurane on oxygenation and shunt fraction during one-lung ventilation. Anesth Analg. 1998 Nov;87(5):1164-9. doi: 10.1097/00000539-199811000-00035. PMID 9806702
- [Result] Xu WY, Wang N, Xu HT, Yuan HB, Sun HJ, Dun CL, Zhou SQ, Zou Z, Shi XY. Effects of sevoflurane and propofol on right ventricular function and pulmonary circulation in patients undergone esophagectomy. Int J Clin Exp Pathol. 2013 Dec 15;7(1):272-9. eCollection 2014. PMID 24427348
- [Result] Voigtsberger S, Lachmann RA, Leutert AC, Schlapfer M, Booy C, Reyes L, Urner M, Schild J, Schimmer RC, Beck-Schimmer B. Sevoflurane ameliorates gas exchange and attenuates lung damage in experimental lipopolysaccharide-induced lung injury. Anesthesiology. 2009 Dec;111(6):1238-48. doi: 10.1097/ALN.0b013e3181bdf857. PMID 19934867
- [Result] Ferrando C, Aguilar G, Piqueras L, Soro M, Moreno J, Belda FJ. Sevoflurane, but not propofol, reduces the lung inflammatory response and improves oxygenation in an acute respiratory distress syndrome model: a randomised laboratory study. Eur J Anaesthesiol. 2013 Aug;30(8):455-63. doi: 10.1097/EJA.0b013e32835f0aa5. PMID 23545542
- [Result] Kellner P, Muller M, Piegeler T, Eugster P, Booy C, Schlapfer M, Beck-Schimmer B. Sevoflurane Abolishes Oxygenation Impairment in a Long-Term Rat Model of Acute Lung Injury. Anesth Analg. 2017 Jan;124(1):194-203. doi: 10.1213/ANE.0000000000001530. PMID 27782948
- [Result] Ma X, Vervoort D. Critical care capacity during the COVID-19 pandemic: Global availability of intensive care beds. J Crit Care. 2020 Aug;58:96-97. doi: 10.1016/j.jcrc.2020.04.012. Epub 2020 Apr 23. No abstract available. PMID 32408107
- [Result] Sylvester JT, Shimoda LA, Aaronson PI, Ward JP. Hypoxic pulmonary vasoconstriction. Physiol Rev. 2012 Jan;92(1):367-520. doi: 10.1152/physrev.00041.2010. PMID 22298659
- [Result] Abbas AE, Fortuin FD, Schiller NB, Appleton CP, Moreno CA, Lester SJ. A simple method for noninvasive estimation of pulmonary vascular resistance. J Am Coll Cardiol. 2003 Mar 19;41(6):1021-7. doi: 10.1016/s0735-1097(02)02973-x. PMID 12651052
- [Result] Lindqvist P, Soderberg S, Gonzalez MC, Tossavainen E, Henein MY. Echocardiography based estimation of pulmonary vascular resistance in patients with pulmonary hypertension: a simultaneous Doppler echocardiography and cardiac catheterization study. Eur J Echocardiogr. 2011 Dec;12(12):961-6. doi: 10.1093/ejechocard/jer222. Epub 2011 Oct 19. PMID 22011836
- [Result] Venkateshvaran A, Hamade J, Kjellstrom B, Lund LH, Manouras A. Doppler estimates of pulmonary vascular resistance to phenotype pulmonary hypertension in heart failure. Int J Cardiovasc Imaging. 2019 Aug;35(8):1465-1472. doi: 10.1007/s10554-019-01591-z. Epub 2019 May 23. PMID 31123846
- [Result] Augustine DX, Coates-Bradshaw LD, Willis J, Harkness A, Ring L, Grapsa J, Coghlan G, Kaye N, Oxborough D, Robinson S, Sandoval J, Rana BS, Siva A, Nihoyannopoulos P, Howard LS, Fox K, Bhattacharyya S, Sharma V, Steeds RP, Mathew T. Echocardiographic assessment of pulmonary hypertension: a guideline protocol from the British Society of Echocardiography. Echo Res Pract. 2018 Sep;5(3):G11-G24. doi: 10.1530/ERP-17-0071. PMID 30012832
- [Result] Walley KR. Use of central venous oxygen saturation to guide therapy. Am J Respir Crit Care Med. 2011 Sep 1;184(5):514-20. doi: 10.1164/rccm.201010-1584CI. PMID 21177882
- [Result] Cruz JC, Metting PJ. Understanding the meaning of the shunt fraction calculation. J Clin Monit. 1987 Apr;3(2):124-34. doi: 10.1007/BF00858361. PMID 3585433